CLINICAL TRIAL: NCT06929091
Title: Ready, Set, Nourish Study
Brief Title: Effect of Prenatal and Postnatal Intervention Strategies on Breastfeeding Outcomes in Women With Excessive Weight (Ready, Set, Nourish Study)
Acronym: RSN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Arkansas Children's Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 298382
Record Dates: First submitted 2025-04-08; First posted 2025-04-16 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Breastfeeding; Dietary Intervention; Milk Expression, Breast
Keywords: Breastfeeding; Human Milk; Obesity; Health Diet
MeSH Terms: conditions — Breast Feeding; Breast Milk Expression; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Lactation support group (Experimental): This group helps researchers compare the effects of the intervention by serving as a baseline for what would happen without ABME technique or a dietary intervention.
  Interventions: Other: Lactation Support
- Lactation Support + Prenatal Intervention group (Experimental): Participants in this group will receive instructions on Antenatal Breast Milk Expression (ABME) and have collection of colostrum before delivery.
  Interventions: Other: Lactation Support and ABME
- Lactation Support + Postnatal Intervention group (Experimental): Participants will receive lactation support and a 5.5-month postpartum dietary program aligned with the Dietary Guidelines for Americans.
  Interventions: Other: Lactation Support and meal plan

INTERVENTIONS:
Other: Lactation Support and ABME — Participants randomized to this group will receive lactation support as group 1. They will also receive education and training (video and handout) on hand expression of colostrum, ABME technique, starting at ~ 37 weeks of gestation. They will have Q&A session with a CLC to address individual concerns and reinforce proper technique. Participants will be asked to perform hand expression 2 times per day for 2-5 minutes, store the colostrum according to the instructions they will receive and bring the sample on the first postnatal study visit.
  Arms: Lactation Support + Prenatal Intervention group
Other: Lactation Support and meal plan — Participants randomized to this group will receive similar lactation support as group 1. They will also receive a 5.5-month dietary program postpartum, designed to align with the Dietary Guidelines for Americans. The plan emphasizes lean proteins, legumes, nuts, whole grains, fruits, vegetables, low-fat dairy, and healthy fats. Up to two daily meals (lunch and dinner) will be delivered as packaged, made-to-order meals. Breakfast items, wraps, and snacks (e.g., shakes) will be prepared by participants using whole foods provided by the facility, with a blender supplied if needed. Additional snacks and items will be given during study visits. Participants will be encouraged to follow the plan consistently, including outside the home, but may have one "flex" day per week to eat outside the plan. Compliance will be monitored with 24-hour recalls and consultations with a nutritionist at each visit.
  Arms: Lactation Support + Postnatal Intervention group
Other: Lactation Support — Participants randomized to this group will receive standard prenatal and postnatal lactation support, including prenatal breastfeeding education with handouts, videos and interaction with certified lactation counselors (CLC), as well as postpartum lactation support as needed by CLCs.
  Arms: Lactation support group

SUMMARY:
This study is about preparing women with excessive weight to have better breastfeeding outcomes. By doing this study, the investigators hope to learn more about how hand expression of breast milk or colostrum during pregnancy can help prepare a mother to breastfeed after she has her baby and about how her diet affects the composition of her breast milk and her baby's growth and development.

DETAILED DESCRIPTION:
The American Academy of Pediatrics recommends exclusive breastfeeding for at least 6 months followed by continued breastfeeding with the introduction of complementary foods as long as desired. When started during the first hour after birth, breastfeeding is more successful. In Arkansas, 74% of infants are breastfed at some point and 24% are exclusively breastfed through 6 months. As such, human milk serves as the primary source of nutrition for many infants. Current research demonstrates lower breastfeeding initiation and shortened duration of breastfeeding in women with obesity. Barriers are present to supporting women with obesity and overweight to successfully breastfeed and meet the breastfeeding recommendations. One barrier is that women with pre-pregnancy obesity have an increased risk of delayed lactogenesis II.

It is unclear what the most effective strategies may be to support women with obesity and overweight to meet their breastfeeding goals. Specifically, there is lack of evidenced-based literature for women with overweight and obesity who want to breastfeed. Findings suggest that targeted interventions in early pregnancy can help ameliorate the effects of obesity and poor breastfeeding initiation as an innovative opportunity to improve breastfeeding rates in this group. Recent research shows that women with overweight and obesity who receive additional support and education to breastfeed from a physician increase their likelihood to initiate breastfeeding. Educational interventions and support, specifically from health professionals tailored towards women with overweight and obesity may improve breastfeeding initiation, exclusivity, and duration.

Antenatal breastmilk expression (ABME) is an innovative technique of colostrum expression in the later weeks of pregnancy (36 weeks to birth) that can be used as a targeted intervention to support women at risk of not breastfeeding or early breastfeeding cessation. ABME starting at 37 weeks gestation has been shown to have the potential to hasten the onset of lactogenesis II, can improve postpartum engorgement, decrease need for supplementation in infants, and improve exclusive breastfeeding duration up to six months postpartum. The limited research on ABME has been mostly in regards to mothers with gestational diabetes and/or for reduction of newborn hypoglycemia. In a recently published systematic review, the findings demonstrated that there is limited evidence and few research studies that have tested the feasibility of antenatal breastmilk expression. Based upon these reviews and the limited evidence from small qualitative studies, more research is needed regarding the efficacy, feasibility, and acceptability of ABME to help women with excessive weight to meet their breastfeeding goals.

Breastfeeding can play a significant role in improving maternal and child outcomes, especially in preventing childhood obesity. Epidemiological and experimental studies support the influence mother's diet in milk composition via several pathways that modulate direct and indirectly certain milk components. Dietary habits, and excessive weight among other factors has been associated with compositional changes in human milk including increased human milk concentrations of leptin, insulin, C-reactive protein, fat, protein and some oligosaccharides. All of these have also been associated with elevated infant fat mass index, even after considering daily human milk volume intakes or adjusting for maternal body mass index and birth weight. In the United States, more than half of women of childbearing age are with excessive weight, which may affect their milk composition and be an early programming of health in later life.

Despite such evidence, no specific dietary recommendations currently exist for lactating women with excessive weight to promote optimal breastfeeding outcomes, human milk composition, infant growth, and infant body composition. In fact, the current report of the Dietary Guidelines for Americans Advisory Committee (2025) pointed to numerous gaps in knowledge that limited their ability to provide strong dietary recommendations for pregnant and lactating women with excessive weight. Therefore, understanding the associations between human milk composition and developmental outcomes can lead to strategies for modifying maternal dietary habits when needed. Considering that most factors happening in the first 1000 days of life represent risk for the development of later childhood obesity are modifiable, a study that will investigate quantitative and qualitative the role of maternal diet on breast milk composition, associate maternal and infant metabolic state and anthropometric characteristics can contribute with evidences to next recommendations for these public.

Hypothesis and/or Specific Aims or Objectives The primary aim of the study is to test whether prenatal and postnatal intervention strategies can impact breastfeeding outcomes for women with excessive weight. The objectives of the study is to test a dietary intervention designed to meet the Dietary Guidelines for Americans and to evaluate whether health care professional education about ABME during pregnancy can improve breastfeeding outcomes and human milk composition in women with overweight or obesity.

The study proposes the hypotheses that in lactating women with excessive weight a dietary intervention during the first 5.5 months postpartum will optimize human milk composition and breastfeeding outcomes. Completion of this research plan will provide evidence-based data for future dietary guidance for lactating women with excessive weight.

The further hypothesize that antenatal breastmilk expression starting ~ 37 weeks gestation will improve breastfeeding outcomes, such as breastfeeding initiation, duration, exclusivity, and decreased delay in lactogenesis II, in women with overweight and obesity.

Outcomes

* Primary: Dietary intervention and ABME interventions will improve breastfeeding outcomes, such as optimizing human milk composition, and breastfeeding initiation and duration, compared to the lactation support group.
* Secondary: Breastfeeding exclusivity up to 6 months, decreased delay in lactogenesis II, and increased breastfeeding self-efficacy, and human milk composition.

ELIGIBILITY:
Inclusion Criteria

* Age 18 or older
* Less than 37 weeks of pregnant with singleton fetus
* Pre-pregnancy excessive weight (Body Mass Index ≥ 25 kg/m2)
* Interested in breastfeeding
* Willing to express colostrum from around 37 weeks of pregnancy if randomized to the prenatal intervention group
* Willing to express human milk for sample collection during a 24-hour period
* Willing to adhere to a meal plan for 5.5 months post-partum if randomized to the postnatal intervention group
* Able to engage in study procedures for the first 24 months postpartum
* Reside in Central Arkansas region Exclusion Criteria
* Pre-existing conditions (e.g. diabetes, hypertension, heart disease, thyroid disorders);
* Use of recreational drugs, tobacco, or 2 or more servings of alcohol per month
* Food allergies, intolerances, or preferences interfering with the meal plan
* Medical history including any contraindication to breastfeeding (medications or supplements incompatible with breastfeeding, substance use)Multiparous pregnancy
* History of breast surgery or radiation
* Congenital defects
* Preeclampsia

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 240 (Estimated)
Dates: Start 2025-11-07 (Actual); Primary Completion 2028-10-01 (Estimated); Study Completion 2029-12-01 (Estimated)

PRIMARY OUTCOMES:
Human Milk composition | From birth to 6 months postpartum
  Human Milk composition will be analyzed from milk samples collected at the postpartum visits (2 weeks, 1, 2, 3, 4, 5, and 6 months). Standardized collection and laboratory procedures described in the study protocol will be followed. Samples will be stored and analyzed at the Arkansas Children's Nutrition Center to evaluate milk composition over time across study groups.
Breastfeeding Initiation | Birth to 2 weeks postpartum
  Breastfeeding initiation (defined as any breastfeeding within the first 24 hours after delivery) will be assessed using standardized Lactation Medical History questionnaire. Data will be obtained at first postpartum study visit, occurring at approximately 2 weeks postpartum. This assessment will provide quantitative data on breastfeeding practice across all study groups.
Breastfeeding Duration | From birth to 6 months
  Breastfeeding duration (measured in cumulative days of any breastfeeding and exclusive breastfeeding) will be assessed using a standardized Lactation Medical History questionnaire. Data will be obtained at all postpartum study visits occurring approximately at 0.5, 1, 2, 3, 4, 5, and 6 months postpartum. These assessments will provide quantitative data on breastfeeding practices across all study groups.

SECONDARY OUTCOMES:
Delay in Onset of Lactogenesis II | From delivery to 1 month postpartum.
  Onset of copious milk secretion (Lactogenesis II) will be assessed by maternal self-report at the first postpartum study visits. Delay in Lactogenesis II will be defined as onset ocurring more than 72 hours after delivery. Data will be collected through the Postnatal Lactation Medical History questionnaire.
Breastfeeding Self-Efficacy Scale- Short | From birth to 2 weeks postpartum.
  Maternal confidence in breastfeeding ability will be evaluated using the Breastfeeding Self-Efficacy Scale-Short Form. The Breastfeeding Self-Efficacy Scale - Short Form measures a mother's confidence in her ability to breastfeed. It consists of 14 items rated on a 5-point Likert scale (1=not at all confident, 2= not very confident, 3=sometimes confident, 4= confident, 5= always confident). Possible range: minimum 14 (if all responses=1) and maximum 70 (if all responses=5). Higher scores (closer to 70) indicate greater breastfeeding self-efficacy (i.e., mother is confident in breastfeeding, more likely to continue breastfeeding and less likely to supplement or wean early). Moderate scores (40-55) indicate variable or developing confidence (i.e., mother may need guidance, and support). Low scores (closer to 14-39) indicate low breastfeeding self-efficacy (i.e., mother may have concerns, or challenges). The questionnaire will be administered at the first postpartum visit (2 weeks).
Breastfeeding Exclusivity up to 6 Months | From birth through 6 months postpartum.
  Exclusive breastfeeding status will be determined through maternal self-report using the Postnatal Lactation Medical History questionnaire. Exclusivity will be defined as no other liquids or solids except for prescribed vitamins or medications given to the infant. Assessments will occur at each postpartum visit ( 0.5, 1, 2, 3, 4, 5, and 6 months).

CONTACTS AND LOCATIONS:
Locations (1):
- Arkansas Children's Nutrition Center, Little Rock, Arkansas, United States

IPD SHARING:
Plan to Share IPD: No
We do not plan to share individual participant data (IPD) from this study. The data will be used in aggregated form only, solely for the purposes of scientific publication and dissemination of the study results. Individual-level data will not be made available to other researchers due to privacy concerns, ethical restrictions, and the terms of the informed consent provided to participants.